CLINICAL TRIAL: NCT03368625
Title: A Phase II Study of Neoadjuvant Stereotactic Radiosurgery for Large Brain Metastases
Brief Title: A Study of Neoadjuvant Stereotactic Radiosurgery for Large Brain Metastases
Acronym: NASRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5689
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Brain Metastases
Keywords: Stereotactic Radiosurgery; Radiation; Surgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Patients with resectable brain mets will receive neoadjuvant stereotactic radiosurgery prior to surgical resection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): Neoadjuvant SRS
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Stereotactic Radiosurgery before surgical resection of brain mets.

SUMMARY:
This study will be a non-randomized phase II trial for patients with one to six brain metastases, at least one of which is appropriate for surgical resection. Upon registration, patients will be assigned to receive neo-adjuvant stereotactic radiosurgery (NASRS).

DETAILED DESCRIPTION:
Recently, a novel treatment strategy for large brain metastases was described whereby lesions appropriate for resection were treated with a single fraction of SRS pre-operatively. In a retrospective analysis, of 51 lesions with a median tumor size of 3 cm, 1-year LC was 86%. This neoadjuvant approach resulted in lower rates of leptomeningeal failure (3 vs. 17%) and symptomatic radiation toxicity (1.5 vs. 14.6 %) compared to a comparative cohort of lesions treated with post-operative cavity boost SRS (POCBS).

Based on promising results, we believe that a prospective trial to establish the value of neoadjuvant SRS (NaSRS) for the treatment of BM appropriate for resection is warranted.

This study will be a non-randomized phase II trial for patients with one to six brain metastases, at least one of which is appropriate for surgical resection. Upon registration, patients will be assigned to receive neo-adjuvant stereotactic radiosurgery (NASRS).

ELIGIBILITY:
Inclusion Criteria:

* Lymphoma, small cell carcinoma, and seminoma are excluded
* A lesion appropriate for resection, not previously treated with SRS. Lesions should be > 2 cm and < 4 cm in largest dimension, and require resection ( e.g. due to mass effect or to obtain a tissue diagnosis). Index lesions will be treated with SRS and surgery, as outlined in the treatment section of the protocol.
* Seen by a neurosurgeon or radiation oncologist and judged to be appropriate for participation in this study, including the ability to tolerate NaSRS, e.g., the ability to lie flat in a stereotactic head frame.
* Any unresected lesions or lesions for which there is no planned immediate resection (non index lesions) must measure < 3.0 cm in maximal extent on the contrasted MRI or CT brain scan obtained ≤ 35 days prior to pre-registration. Unresected lesions will be treated with SRS as outlined in the treatment section of the protocol. .
* ECOG ≤ 2
* MRI confirmed 1-6 lesions, one of which is the index lesion. Each non-index lesion (up to 5) must measure ≤ 3.0 cm in maximal extent on contrasted MRI scan, and not otherwise require resection.

Note: The pre-registration MRI may be obtained ≤ 35 days prior to enrolment.

Exclusion Criteria:

* Treatment plan respecting normal tissue tolerances using dose fractionation specified within the protocol cannot be achieved.
* pregnancy
* Prior cranial radiotherapy targeting the index lesion, or any prior WBRT.
* Inability to complete a MRI with contrast of the head, or a known allergy to gadolinium.
* Cytotoxic Chemotherapy within 7 days prior to SRS (molecularly targeted therapies , including immune-modulatory drugs, can be given within seven days of SRS at the discretion of the treating physician)
* Metastatic germ cell tumor, small cell carcinoma, or lymphoma or any primary brain tumor
* Imaging Findings:

  * Widespread definitive leptomeningeal metastasis.
  * A brain metastasis that is located ≤ 2 mm of the optic chiasm
  * Evidence of midline shift
  * Fourth ventricular narrowing, concerning for hydrocephalus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiation toxicity | 1 year
  The rate at 1 year of symptomatic (≥grade 2) radiation toxicity

SECONDARY OUTCOMES:
local control | 1 year
  1-year local control (PR+CR) of the index lesion resulting from NaSRS
leptomeningeal disease | 1 year
  1-year rates of leptomeningeal disease
Survival | 5 years
  Median survival
progression-free survival | 2 years
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Shultz, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- University Health Network, Toronto, Ontario, Canada
- Charité Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Higazy R, Li D, Lau R, Millar BA, Laperriere N, Berlin A, Conrad T, Gutierrez-Valencia E, Zadeh G, Bernstein M, Kalyvas A, Spears J, Zips D, Vajkoczy P, Senger C, Acker G, Kongkham P, Shultz DB. Neoadjuvant Stereotactic Radiosurgery for Large Brain Metastases: An International, Multicenter, Single-Arm Phase II Trial. Neurosurgery. 2025 Apr 14;97(4):793-800. doi: 10.1227/neu.0000000000003451. PMID 40227031